CLINICAL TRIAL: NCT03677765
Title: A Prospective Non-inferiority Trial on Complications Related to Ultrasonography-guided Subclavian Venous Catheterization: Supraclavicular Versus Infraclavicular Approach
Brief Title: Comparisons of Complications Related to Two Approaches of Ultrasonography-guided Subclavian Venous Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: US_SVC: SC vs IC
Record Dates: First submitted 2018-09-09; First posted 2018-09-19 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Complication of Treatment; Catheterization
Keywords: subclavian venous catheterization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infraclavicular group (Active Comparator): In the infraclavicular group, subclavian venous catheterization using ultrasonography is performed beneath the clavicle.
  Interventions: Procedure: Supra- vs Infraclavicular approach using ultrasonography
- Supraclavicular group (Active Comparator): In the supraclavicular group, subclavian venous catheterization using ultrasonography is performed over the clavicle.
  Interventions: Procedure: Supra- vs Infraclavicular approach using ultrasonography

INTERVENTIONS:
Procedure: Supra- vs Infraclavicular approach using ultrasonography — In the supraclavicular group, subclavian venous catheterization using ultrasonography is performed beneath the clavicle. Meanwhile, in the infraclavicular group, subclavian venous catheterization using ultrasonography is performed over the clavicle.

SUMMARY:
For performing subclavian venous catheterization, two approaches (supraclavicular and infraclavicular) have been used successfully in various clinical practice. However, there remains controversy concerning which approach is safer and causes less complications during ultrasonography-guided subclavian venous catheterization. In this context, the investigators sought to compare supraclavicular approach with infraclavicular approach in terms of post-procedural complications during ultrasonography-guided subclavian venous catheterization.

ELIGIBILITY:
Inclusion Criteria:

* patients who require subclavian venous catheterization
* adult patients aged 20-79

Exclusion Criteria:

* patient's refusal
* patients with contraindication of subclavian venous catheterization (skin infection at puncture site, tumor or thrombus in the course of subclavian vein, vegetation at tricuspid valve, patients on anticoagulation)
* patients with chemoport or pacemaker in subclavian vein
* patients with right-sided breast cancer operation or with right-sided pneumonectomy

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
the overall incidence of complications | intraoperatively to 1 hour after the admission of ICU
  The overall incidence of complications will be expressed as the sum of incidences of complications which occurred during subclavian venous catheterization including arterial puncture, hematoma formation, pneumothorax, hemothorax, and malposition of catheter. Arterial puncture, hematoma formation, and malposition of catheter will be evaluated with ultrasonography, and pneumothorax and hemothorax will be evaluated by chest radiography.

SECONDARY OUTCOMES:
the first-pass success rate | intraoperatively
  The first-pass success was defined as successful catheterization on a single attempt in all stages of catheterization.
the number of needling for venipuncture | intraoperatively
  The number of needling for venipuncture was defined as the amount of needling for successful subclavian venous puncture.
Total time for venipuncture | intraoperatively
  Total time for venipuncture was defined as the amount of time which took for successful subclavian venous puncture.

CONTACTS AND LOCATIONS:
Overall Officials: Hee-pyoung Park, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim YJ, Ma S, Yoon HK, Lee HC, Park HP, Oh H. Supraclavicular versus infraclavicular approach for ultrasound-guided right subclavian venous catheterisation: a randomised controlled non-inferiority trial. Anaesthesia. 2022 Jan;77(1):59-65. doi: 10.1111/anae.15525. Epub 2021 Jul 6. PMID 34231204